CLINICAL TRIAL: NCT03365713
Title: Global Excellence in COPD Outcomes: Implementation and Effectiveness of COPD Case-Finding in Low and Middle Income Countries
Brief Title: GECo: Implementation and Effectiveness of COPD Case-Finding in Low and Middle Income Countries
Acronym: GECo1
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Collaborators: Johns Hopkins University (Other); Universidad Peruana Cayetano Heredia (Other); Asociacion Benefica Prisma (Other); Makerere University (Other); University of York (Other); Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Responsible Party: Sponsor
Other Study IDs: 16/0630_CF
Record Dates: First submitted 2017-11-17; First posted 2017-12-07 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Spirometry; COPD Diagnosis; PEF; Case Finding; LMIC
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will test how well short questionnaires, with and without a simple breathing test called 'peak flow', can identify people with COPD compared to the gold-standard diagnostic test called spirometry. We will test this in 10,500 people from three low- and middle-income countries, namely Nepal, Peru and Uganda. We will also examine the feasibility of implementing our case-finding intervention at scale.

DETAILED DESCRIPTION:
The investigators will determine whether case-finding for COPD can be facilitated using 5-item questionnaires with and without a measurement of Peak-Flow. The investigators hypothesise that 5-item questionnaires will be a valid case-finding tool for COPD in LMIC and will be acceptable and feasible for use in these settings.

1. Clinical Aim: Determine the diagnostic accuracy of the case-finding questionnaires with and without PEF.
2. Implementation Aim: Assess the appropriateness, acceptability and feasibility of using questionnaires and PEF to identify COPD cases from the perspective of local community members, community health workers, local health centre physicians and ministries of health.

The design of the intervention will be informed by formative work prior to commencement of the main study.

Study fieldworkers will enroll and screen a randomly-selected age- and sex-stratified population sample of adults aged ≥40 years; a total of 10,500 between the following three countries in the catchment areas of existing community census areas in Bhaktapur (Nepal), Lima (Peru), and Nakaseke (Uganda).

The investigators will report the sensitivity, specificity and positive predictive value of the case-finding questionnaire, with and without PEF, in relation to a gold standard COPD diagnosis made at spirometry (post-bronchodilator FEV1/VC ratio <LLN, with a history of significant respiratory exposure to tobacco smoke or biomass). The investigators will construct ROC curves to visualise trade-offs in sensitivity and specificity across a range of questionnaire cut off values.

The investigators will also examine the feasibility of implementing a 5 item questionnaire +/- PEF intervention at scale.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged ≥40 years
* Full-time resident in the area (living in area > 6 months)
* Able to perform adequate quality spirometry
* Capable of providing informed consent

Exclusion Criteria:

* Pregnancy (self-reported)
* Currently has active pulmonary TB or is taking medications for pulmonary TB

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A randomly-selected age- and sex-stratified population sample of adults aged ≥40 years; a total of 10,500 will be recruited from the following three countries in the catchment areas of existing community census areas, in Bhaktapur (Nepal), Lima (Peru), and Nakaseke (Uganda).
Sampling Method: Probability Sample
Enrollment: 10709 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

PRIMARY OUTCOMES:
Sensitivity, Specificity and Positive Predictive Value of Simple Case Finding tools | 12 months
  Sensitivity, Specificity and Positive Predictive Value of the case-finding questionnaires with and without peak-expiratory flow (PEF), compared to spirometry.

SECONDARY OUTCOMES:
Process Evaluation - Actual number of participants recruited against target. | 12 months
  Total number of participants successfully recruited into the study against the target figure determined by the power calculations.
Fidelity - Spirometry Quality Control Failures | 12 months
  Extent to which delivery adheres to the protocol developed. Spirometry delivery - Only tests which meet both acceptability and repeatability criteria as per ERS/ATS (European Respiratory Society / American Thoracic Society) guidelines will be accepted.
  Spirometry interpretation - All Spirometry preformed will be over-read locally, and a proportion (see below) will be over-read centrally. Two separate researchers, at each site, adequately trained in both spirometry delivery and interpretation will separately perform interpretation of all spriometry carried out in the field, to ensure correct interpretation in relation to a gold standard COPD diagnosis made at spirometry (post-bronchodilator FEV1/VC ratio <LLN, with a history of significant respiratory exposure to tobacco smoke or biomass) . Of these, 10% will be over-read centrally by the principal investigators to ensure quality assurance.
Fidelity - Proportion of Questionnaires with Missing Data Fields | 12 months
  Extent to which delivery adheres to the protocol developed. The investigators will report the proportion of incomplete questionnaires (any questionnaires with one or more missing data fields) in total and at each individual site.
Health Economics | 12 months
  Health-related productivity costs measured as hours of lost work from COPD and related symptoms.
  Inequalities in productivity costs according to illness severity and wealth status.

CONTACTS AND LOCATIONS:
Overall Officials: John Hurst, PhD FRCP, Principal Investigator — University College, London
Locations (3):
- Institute of Medicine, Kathmandu, Nepal
- Universidad Peruana Cayetano Heredia, Lima, Peru
- Makerere University Lung Institute, Makerere, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Robertson NM, Siddharthan T, Pollard SL, Alupo P, Flores-Flores O, Rykiel NA, Romani ED, Ascencio-Dias I, Kirenga B, Checkley W, Hurst JR, Quaderi S; GECo Investigators. Development and Validity Assessment of a Chronic Obstructive Pulmonary Disease Knowledge Questionnaire in Low- and Middle-Income Countries. Ann Am Thorac Soc. 2021 Aug;18(8):1298-1305. doi: 10.1513/AnnalsATS.202007-884OC. PMID 33476252
- [Derived] Siddharthan T, Pollard SL, Quaderi SA, Mirelman AJ, Cardenas MK, Kirenga B, Rykiel NA, Miranda JJ, Shrestha L, Chandyo RK, Cattamanchi A, Michie S, Barber J, Checkley W, Hurst JR; GECo Study Investigators. Effectiveness-implementation of COPD case finding and self-management action plans in low- and middle-income countries: global excellence in COPD outcomes (GECo) study protocol. Trials. 2018 Oct 19;19(1):571. doi: 10.1186/s13063-018-2909-8. PMID 30340648
- See also: The Johns Hopkins Center for Global NCD Research and Training — https://www.globalncd.org/
- See also: Trial Twitter account - @COPDGECo — https://twitter.com/copdgeco?lang=en